CLINICAL TRIAL: NCT03567824
Title: A Phase 2 Open Label Study of Magnesium L-Lactate Dihydrate (MLD10) 10 mEq Extended-Release Caplets Administered BID for the Treatment of Hypomagnesemic Patients With Type 2 Diabetes Mellitus Followed by a Blinded Random Off Phase
Brief Title: MLD10 for the Treatment of Hypomagnesemic Patients With Type 2 Diabetes Mellitus
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Pharmalyte Solutions LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MLD 10-003
Record Dates: First submitted 2018-05-18; First posted 2018-06-26 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Hypomagnesemia in Type 2 Diabetic Patients

STUDY DESIGN:
Intervention Model Description: All subjects will be treated open label for the first 3 months on study, then randomized to receive either active or placebo for an additional 3 months.
Who Masked: Participant, Investigator
Masking Description: The second phase of the study where subjects are randomized to either active or placebo will be blinded to both participant and investigator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Open label phase (Experimental): MLD10 (magnesium l-lactate dihydrate) 10mEq extended release caplets BID for three months, all subjects.
  Interventions: Drug: Magnesium L-lactate dihydrate
- Random off phase (Other): MLD10 (magnesium l-lactate dihydrate) 10mEq extended release caplets BID for three months or Placebo
  Interventions: Drug: Magnesium L-lactate dihydrate; Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Magnesium L-lactate dihydrate — Magnesium L-lactate dihydrate 10 mEq extended release caplets
  Other Names: MLD10
Drug: Placebo Oral Tablet — Placebo will have the same appearance, taste, odor and mode of administration as MLD10.
  Arms: Random off phase

SUMMARY:
To determine the effect of MLD10 (magnesium L-lactate dihydrate extended-release caplets) 10 mEq BID on serum magnesium in Type 2 diabetic patients with hypomagnesemia.

ELIGIBILITY:
Inclusion Criteria:

* Females and males with Type 2 diabetes mellitus
* Body Mass Index between 18 to 40 kg/m2, inclusive, at Screening
* Hypomagnesemia defined as serum magnesium ≤ 1.5 mg/dL at Screening
* Females must be non-pregnant, non-lactating, and have a negative serum pregnancy test before enrollment.

Exclusion Criteria:

* History of clinically significant GI, renal, hepatic, neurologic, hematologic, endocrine other than Type 2 diabetes mellitus, oncologic, pulmonary, immunologic, psychiatric, or cardiovascular disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in Serum Magnesium Concentration | Three months after the initiation of treatment and then at 3 months after the start of the random off phase.
  Change from baseline in serum magnesium concentration.

SECONDARY OUTCOMES:
Change in Serum Magnesium Concentration. | At 1 and 2 months after the initiation of treatment.
  Change from baseline in serum magnesium concentration.
Change in Fasting Blood Glucose | Three months after the initiation of treatment and then at 3 months after the start of the random off phase.
  Change from baseline in fasting blood glucose.
Change in Insulin Sensitivity | Three months after the initiation of treatment and then at 3 months after the start of the random off phase.
  Change from baseline in insulin sensitivity.
Change in Insulin Resistance | Three months after the initiation of treatment and then at 3 months after the start of the random off phase.
  Change from baseline in insulin resistance.
Change in HbA1c | Three months after the initiation of treatment and then at 3 months after the start of the random off phase.
  Change from baseline in HbA1c.

IPD SHARING:
Plan to Share IPD: Undecided